CLINICAL TRIAL: NCT05709418
Title: Intensiv støtte i Matematikk for Elever Som er i Risiko for å Utvikle Matematikkvansker
Brief Title: Intervention for Low-performing First Graders in Mathematics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ostfold University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OstfoldUC
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Mathematics Disorder
MeSH Terms: conditions — Dyscalculia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mathematics intervention (Experimental): Low-performing children get targeted support with a scripted intervention
  Interventions: Behavioral: Intensiv support for first graders in Norway
- Control group (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Intensiv support for first graders in Norway — Intervention targeting early numeracy skills that are known to be important for mathematical development, focusing on counting skills, counting strategies, number knowledge, word problem solving and basic understanding of addition and subtraction
  Arms: Mathematics intervention

SUMMARY:
The aim of this study is to investigate the effect of an intervention program for low-performing first graders in mathematics. .

DETAILED DESCRIPTION:
There were sent a request to a school in the central of East-Norway to participate. The principal answered yes, and then asked the teachers at first grade if they would like to participate. The teachers were positive to the study, and therefore the students and parents were asked to participate. It was total 74 students and 54 of them accepted to participate in the study. The inclusion criteria of the study is that the participants talks and understand Norwegian approximate fluently. In this study that means one participant was excluded.

The study will use a design of randomized control trial (RCT) where the population of 53 students will be doing av screening-test. After the screening 20% of the lowest-performance will make up the sample and they will be departed in a clinical-group and a control-group. These students will then be tested with Test of Basic Arithmetic and Numeracy, the Norwegian test called Arithmetic fact-test, the vocabulary and calculation tasks from Wechsler Intelligence Scale for Children - Fifth Edition and Ravens colored progressive matrices. The randomization will be conduct using randomize.org and the parents will get information about which group their child will participate in. The intervention are eight week long with 4 lessons per week. Each lesson are about 45-50 minutes long. The start of the intervention will be in week 42, 2022 and end in week 49, 2022. The intervention-group will follow an intervention conducting elements from an education program called "ThinkMath" and self-developed tasks. The control-group will follow ordinary classroom-lessons. After ended intervention-period the students will be tested with the same test-battery as were used in front of the start point.

ELIGIBILITY:
Inclusion Criteria: Performing under the cut off score of a screening tool for first graders, i.e. 20th percentile

-

Exclusion Criteria:

* not proficient Norwegian language skills

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number knowledge | 10 weeks
  Number knowledge measured by digit comparison, number reading and number recognition (numerical knowledge) - both orally and written presented. Higher score indicates better result.
Arithmetic fluency 1-10 with Test of Basic Arithmetic and Numeracy, the Norwegian test called Arithmetic fact-test and a digital test created by University of Oslo. | 10 weeks
  Arithmetic fluency in the number area 1-10. Higher score indicates better result.

SECONDARY OUTCOMES:
Word problem solving from Wechsler Intelligence Scale for Children - Fifth Edition | 10 weeks
  Word problem solving presented orally. Minimum score 0, maximum 34. Higher score indicates better result.

OTHER OUTCOMES:
Non-verbal IQ Raven | 10 weeks
  Raven's colored matrices. Minimum score 0, maximum 36. Higher score indicates better result.
Vocubulary from Wechsler Intelligence Scale for Children - Fifth Edition | 10 weeks
  Vocabulary assessment. Minimum score 0, maximum 54. Higher score indicates better result.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Lopez-Pedersen, Phd, Study Chair — Østfold University College
Locations (1):
- Østfold University College, Halden, Norway

IPD SHARING:
Plan to Share IPD: No